CLINICAL TRIAL: NCT02796924
Title: The Efficacy of Transcranial Magnetic Stimulation in the Treatment of Non-epileptic Seizures
Brief Title: Treating Non-epileptic Seizures Using Magnetic Brain Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2016:039
Record Dates: First submitted 2016-06-03; First posted 2016-06-13 (Estimated); Results first posted 2020-09-30 (Actual); Last update posted 2020-09-30 (Actual); Status verified 2020-03

CONDITIONS: Nonepileptic Seizures
Keywords: Psychogenic Non-Epileptic Seizure; Transcranial Magnetic Stimulation; Brain Stimulation
MeSH Terms: conditions — Seizures; Psychogenic Nonepileptic Seizures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients (Experimental): 30 sessions of high-frequency (20Hz) repetitive stimulation applied over the right temporal-parietal junction in patients with psychogenic non-epileptic seizures using a MagStim Rapid2 Transcranial Magnetic Simulation machine.
  Interventions: Device: MagStim Rapid2 Transcranial Magnetic Simulation

INTERVENTIONS:
Device: MagStim Rapid2 Transcranial Magnetic Simulation — A non-invasive method of brain stimulation

SUMMARY:
The purpose of this study is to investigate the feasibility of using repetitive transcranial magnetic stimulation (rTMS) - a form of non-invasive brain stimulation - to decrease the frequency of psychogenic non-epileptic seizure (PNES) episodes in patients with PNES.

DETAILED DESCRIPTION:
This study is an open label pilot study that aims to recruit 15 individuals with diagnosed PNES to investigate the feasibility of using repetitive transcranial magnetic stimulation (rTMS) to decreasing the frequency of psychogenic non-epileptic seizure (PNES) episodes. rTMS is a non-invasive method of brain stimulation that uses rapid magnetic pulses applied over the scalp to active neurons in a specified target location of the brain.

Electronic as well as paper-and-pencil questionnaires will be used to asses patient's psychiatric symptoms and functional impairment both before and after treatment to monitor symptom-changes.Treatment will consist of daily sessions of high frequency (20 Hz) rTMS applied over the right temporoparietal junction (TPJ) of the cerebral cortex. Patients will receive two sessions per day for 15 consecutive weekdays. Each session will take approximately 20 minutes to complete.

Results of the questionnaires will be analyzed to determine the effect of the treatment on PNES episodes and functional impairment. As a pilot study, this research will be used to evaluate the effect size and the feasibility of a more definitive project in the future. Both patient response and tolerability to rTMS will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed Psychogenic Non-Epileptic Seizures

Exclusion Criteria:

* Evidence of previous or comorbid epileptic seizures
* Major comorbid neurological diseases
* Currently taking medications that are known to reduce seizure-threshold
* Currently pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2019-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mandana Modirrousta, MD PhD FRCPC, Principal Investigator — University of Manitoba

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patients
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Patients
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.9 (8.0)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Female | 7
  Gender: Male | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 1
  Unknown or Not Reported | 7
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 10
Number of weekly seizure-events [Mean (Standard Deviation); unit: events] | 8.1 (6.0)

OUTCOME MEASURES:

1. Primary Outcome: Number of Weekly Psychogenic Non-epileptic Seizure-events
Description: Number of weekly seizure-events recorded using seizure logs.
Time Frame: One week and three months post-rTMS treatment
Measure: Mean (Standard Deviation); unit: events
Arm/Group | Patients
Number analyzed (Participants) | 10
events
  One week post-rTMS | 6.9 (15.5)
  Three months post-rTMS | 5.3 (9.6)

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | Patients
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 9/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients (N=10)
Headache (Nervous system disorders) | 6 (6)
Fatigue (Nervous system disorders) | 4 (4)
Vivid dreams (Nervous system disorders) | 4 (4)
Pain (Nervous system disorders) | 1 (1) — Pain at site of stimulation
Nausea (Nervous system disorders) | 1 (1)
Migraine (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-06): https://cdn.clinicaltrials.gov/large-docs/24/NCT02796924/Prot_SAP_000.pdf